CLINICAL TRIAL: NCT01169740
Title: Comparison of Transcutaneous or Laboratory Measurement of Bilirubin in the Newborn
Brief Title: Transcutaneous Measurement of Jaundice in the Newborn
Acronym: TcBili
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Bilirubin 2010/413
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hyperbilirubinemia, Neonatal; Jaundice, Neonatal
Keywords: Hyperbilirubinemia; Neonatal; Serum bilirubin; Transcutaneous bilirubin; Skin color
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal; Hyperbilirubinemia | interventions — Blood Specimen Collection; Skin Pigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonatal jaundice: Infants born between July 1st 2010 and July 31st 2010 and admitted to normal newborn nursery
  Interventions: Procedure: Measurement of bilirubin in blood and skin color

INTERVENTIONS:
Procedure: Measurement of bilirubin in blood and skin color — Blood sampling and analysis, measurement of skin color by transcutaneous bilirubinometry
  Other Names: Diagnosis of jaundice

SUMMARY:
Prospective comparison of measurement of bilirubin in jaundiced newborns by a transcutaneous device (bilirubinometer) and laboratory analysis of blood samples.

We hypothesise that correlation of the two measurements depend on bilirubin level, gestational age as well as postnatal age.

DETAILED DESCRIPTION:
Whenever a blood sample is drawn for measurement of bilirubin in a newborn, a transcutaneous measurement of skin yellow color will be made. Such measurements will also be included in all infants when a CRP-test (blood sample for C-reactive protein) has been ordered, as well as in connection with the routine blood sampling for metabolic screening. Only infants where parents have given written consent for their infant will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infant admitted to normal newborn nursery

Exclusion Criteria:

* Informed consent not obtained

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants admitted to normal newborn nursery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Comparison of transcutaneous bilirubin (skin color, TcB) and bilirubin measured in a blood sample (TsB) | 12 months
  To have statistical strength for comparison of the two tests between 1500 and 2000 patients are needed

SECONDARY OUTCOMES:
Differences in TcB measured at the forehead or at the sternum | 12 months
  To have statistical strength for comparison of the two tests between 1500 and 2000 patients are needed

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Videm, MD, PhD, Study Chair — Norwegian University of Science and Technology, Instititue director
Locations (1):
- St. Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No